CLINICAL TRIAL: NCT04821466
Title: The Use of Virtual Reality for Symptom Control and Wellbeing in Palliative Care and Oncology Patients
Brief Title: VR for Symptom Control and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021.RCHT.07
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Oncology; End Stage Cancer; Palliative Care; Hematologic Malignancy
Keywords: Virtual Reality
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Cohort interrupted time series study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Headset (Experimental): VR headset, programmed with a selection of 7 wellbeing programs to identify if use will improve participants wellbeing
  Interventions: Device: Virtual Reality Headset to provide a Virtual Reality Experience

INTERVENTIONS:
Device: Virtual Reality Headset to provide a Virtual Reality Experience — Participants will utilise a Virtual Reality experience for distraction therapy via a Virtual reality headset. Participants will wear the Virtual reality headset to be immersed in a multimedia experience.

SUMMARY:
To investigate the effect that a Virtual Reality experience can have on patient symptoms and wellbeing for palliative care and oncology inpatients

ELIGIBILITY:
Inclusion criteria

* > 18 years of age
* Inpatient at RCHT know to the palliative care team
* Able to consent
* Able to speak and understand the English language
* Able to use the virtual reality system
* Able to complete ESAS-r Questionnaire

Exclusion criteria

* <18 years of age
* Patient unable to consent
* Patient unable to speak English
* Unable to use the virtual reality system (e.g. visually impaired)
* Known Epilepsy or seizures or suspected predisposition to seizures (e.g. Brain metastasis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
ESAS-r Quality of Life Scores | Time 0 & Time 60 minutes
  Change in ESAS-r QoL score between start and finish of Virtual Reality experience. 0 = No symptoms to 10 = Worst Symptom

SECONDARY OUTCOMES:
Quantitative clinician experience of VR intervention | Time 60 minutes
  Clinician score of patient experience using Virtual Reality intervention for symptoms and wellbeing between 0 (negative) and 10 (positive)
Quantitative clinician experience of VR intervention | Time 60 minutes
  Patient score of experience using Virtual Reality intervention for symptoms and wellbeing between 0 (negative) and 10 (positive)

OTHER OUTCOMES:
Qualitative patient experience of VR interventions | Time 60 minutes
  Patients to answer: Were there any negative side effects of the VR session?
Repeat VR experiences | 12 Months
  ESAS-r QoL Scores (0 to 10) will be collected each time a patient uses the experience to consider the effect repeat exposure has on wellbeing and symptoms. 0 = No symptoms to 10 = Worst Symptom

CONTACTS AND LOCATIONS:
Overall Officials: Niall O Moon, BMBCh, Principal Investigator — Doctor
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share patient data

REFERENCES:
- [Derived] Moon NO, Henstridge-Blows JR, Sprecher EA, Thomas E, Byfield A, McGrane J. 'Godrevy Project': virtual reality for symptom control and well-being in oncology and palliative care - a non-randomised pre-post interventional trial. BMJ Oncol. 2023 Dec 18;2(1):e000160. doi: 10.1136/bmjonc-2023-000160. eCollection 2023. PMID 39886490